CLINICAL TRIAL: NCT01857791
Title: Efficacy of a Clinic-based, Multi- Disciplinary, Pediatric Weight Management Program
Acronym: REWARD Teens
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Vermont (Other)
Responsible Party: Principal Investigator, Connie Tompkins, PhD, Assistant Professor, University of Vermont
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M11-083
Record Dates: First submitted 2013-05-15; First posted 2013-05-20 (Estimated); Last update posted 2015-09-10 (Estimated); Status verified 2015-09

CONDITIONS: Body Weight Changes
MeSH Terms: conditions — Body Weight Changes | interventions — Behavior Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- multidisciplinary, behavior modification (Experimental)
  Interventions: Behavioral: multidisciplinary, behavior modification

INTERVENTIONS:
Behavioral: multidisciplinary, behavior modification

SUMMARY:
Childhood obesity has more than tripled in the past 30 years. From 1980 to 2008, the prevalence of obesity among adolescents aged 12 to 18 years, increased from 5.0% to 18.1%.1 Although several pediatric weight management programs are available, access to these programs may not always be possible.

The proposed study will be an ongoing research program with approximately 40 children ages 12-18 years enrolled into the study over a year. All study participants will participate in a baseline evaluation which will include body composition measures, aerobic testing, as well as nutrition and physical activity questionnaires. Study participants will be assigned to the clinic-based group. The clinic- based group will participate in a 12-week multi-disciplinary weight management program. All study participants will then participate in a 12-week follow-up evaluation similar to the baseline visit. New participants will be enrolled every 12 weeks. Every 12 weeks, active participants (those that have completed a minimum of 12 weeks) will have the option to continue in the program or, discontinue their active participation in the program and enroll into the maintenance phase which will consist of measures only every 12 weeks.

The objective of the proposed study includes examining the efficacy of the clinic-based, multi-disciplinary, pediatric weight management program.

ELIGIBILITY:
Inclusion Criteria:

* Phone screening
* Approval to participate in a weight management program from the child's pediatrician
* Children between the ages of 12 and 18 years
* Children overweight (>85th-<95th BMI percentile) or obese (>95th BMI percentile)

Exclusion Criteria:

* Children with evidence of significant cardiovascular disease or cardiac arrhythmias
* Children with liver disease
* Children on chronic use of medications including diuretics, steroids and adrenergic-stimulating agents
* Children with emotional problems such as clinical depression or other diagnosed psychological condition and currently use prescription medication for psychological conditions
* Children with evidence of family and/or medical neglect or physical, mental or sexual child abuse

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2011-01; Primary Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
weight loss | 12 weeks
  Body weight will be measured at baseline and at 12-weeks. Mean percentage weight change will be assessed following the 12-week intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Vermont, Burlington, Vermont, United States